CLINICAL TRIAL: NCT01342042
Title: The Safety, Preliminary Pharmacodynamics and Pharmacokinetics Study of rExenatide-4 in Chinese T2DM
Brief Title: The Safety,Preliminary Pharmacodynamics and Pharmacokinetics Study of rExenatide-4 in Chinese Type 2 Diabetes Mellitus
Acronym: SPPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other); Peking University First Hospital (Other)
Responsible Party: CSPC ZhongQi Pharmaceutical Technology Co., Ltd., CSPC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC/PRO-rE4/IIa-04
Record Dates: First submitted 2011-04-23; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; rRE-4; exenatide; metformin; CSPC ZhongQi
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Biological: rExenatide-4
- exenatide-4 (Active Comparator)
  Interventions: Biological: rExenatide-4

INTERVENTIONS:
Biological: rExenatide-4 — This protein of 39 amino acids has been isolated from the venom of the lizard Heloderma suspectum (Gila monster) (Eng et al, 1992). A mammalian homolog does not seem to exist (Pohl and Wank, 1998). Exendin-4 shares 53 % identity at the amino acid level with that of the mammalian hormone GLP-1 [glucagon-like peptide-1] (Chen and Drucker, 1997). Exendin-4 is encoded within a prohormone that is distinct from the prohormone encoding glucagon. Using transgenic mice expressing exendin-4, Adatia et al (2002) have shown that mammalian cells process the lizard prohormone in endocrine and nonendocrine cell types in vitro and in murine tissues in vivo.

SUMMARY:
This research is randomized, controlled trial. 36 Chinese subjects with Type 2 Diabetes Mellitus will take part in the trial.

Subjects will randomly enter into one of three groups, administration daily twice, the period of is 84 days treatment. Subjects should be in hospital for pharmacokinetic studies in 1 d~ 8d, 30 d (if necessary)and 84 d, during 9 d ~ 83 d outpatient follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 75 years with T2DM in China;
2. HbA1c of 7% to 13%;
3. negative pregnancy test in females, all subjects have no family planning during the test and after the end within 3 months.

Exclusion Criteria:

1. HBsAg, HCV, HIV and syphilis test was positive;
2. any time FBG <6.1 or> 14.0 mmol / L in the morning;
3. Renal function: eGFR <60 mL / min ;
4. TG> 5mmol / L;
5. Pancreatitis, cholecystitis, gallstones and other gastrointestinal diseases;
6. Ischemic heart disease, heart failure, stroke or peripheral vascular disease;
7. Pregnancy and breast-feeding women;
8. Patients requiring insulin treatment;
9. Have medical history of hypoglycemia;
10. Have a clear history of allergic patients;
11. Patients addicted to alcohol and tobacco.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To compare treatment arms in terms of change from baseline to endpoint in HbA1c | 12 Weeks
  To observe and compare the differences in pharmacokinetic parameters with the reatment of rE-4, adding metformin to rE-4 and exenatide, To compare treatment arms in terms of change from baseline to endpoint in HbA1c

SECONDARY OUTCOMES:
To compare treatment arms in terms of change from baseline to endpoint in GA | 12 Weeks
To compare treatment arms in terms of change from baseline to endpoint in fasting serum glucose | 12 Weeks
To compare treatment arms in terms of change from baseline to endpoint in postprandial blood glucose 2-hour | 12 weeks
To compare treatment arms in terms of change from baseline to endpoint in body weight | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cui Yi min, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Y, Xu B, Zhu L, Lou K, Chen Y, Zhao X, Wang Q, Xu L, Guo X, Ji L, Cui Y, Fang Y. Pharmacokinetics and Preliminary Pharmacodynamics of Single- and Multiple-dose Lyophilized Recombinant Glucagon-like Peptide-1 Receptor Agonist (rE-4) in Chinese Patients with Type 2 Diabetes Mellitus. Clin Drug Investig. 2017 Dec;37(12):1107-1115. doi: 10.1007/s40261-017-0569-1. PMID 28932995